CLINICAL TRIAL: NCT07225881
Title: Efficacy of a Multi-level Intervention Designed to Promote Adherence to WCRF/AICR Dietary Guidelines for Cancer Prevention
Brief Title: Eatwell Clinical Trial (R01)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Meghan Butryn, Professor, Department of Psychological and Brain Sciences, Drexel University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01CA288323 (NIH); R01CA288323 (NIH)
Record Dates: First submitted 2025-10-31; First posted 2025-11-10 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Cancer Prevention; Dietary Guidelines

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eatwell Condition (Experimental): Index participant and household members receive Eatwell intervention
  Interventions: Behavioral: Eatwell
- Comparison Condition (Active Comparator): Index participants receive nutrition education sessions; household members receive no intervention contact
  Interventions: Other: Nutrition Education Control Group

INTERVENTIONS:
Behavioral: Eatwell — The Eatwell intervention content is focused on helping participants make healthier grocery shopping decisions, eat at home more often to take advantage of the optimal defaults present there, and learn how to navigate temptation when eating away from home. The intervention itself involves nutrition education, self-regulation, motivation, and household support. In total, it will last 18 months; index participants will attend 12 workshop sessions that are 90 minutes each. Each workshop session will include approximately 12-16 index participants. The first four sessions will be held weekly in Month 1, and subsequent sessions decrease in frequency. Each index participant will have one enrolled household member who will be asked to join four workshop sessions in a support role: sessions 3, 4, 7, and 10. In these four sessions, household members will receive education about WCRF/AIRC recommendations and training in how to provide instrumental and emotional support to index participants.
  Arms: Eatwell Condition
Other: Nutrition Education Control Group — In the control condition, index participants will receive nutrition education in a series of 12 workshop sessions, following the same schedule as participants in the Eatwell condition. All of the content described under the "nutrition education" component of the Eatwell intervention will be provided. The educational material will be delivered with greater detail and with additional in-session activities, as greater time is devoted to education in the control vs. experimental condition. Participants also will receive monthly educational email messages reiterating key ideas from workshops.
  Specialized content and activities related to self-regulation and motivation will not be provided in the control condition. If an index participant is randomized to the control condition, their designated household member will have no intervention involvement and will only complete assessments.
  Arms: Comparison Condition

SUMMARY:
Cancer is a leading cause of death and will affect many people in their lifetimes. Organizations such as the American Cancer Society and the World Cancer Research Fund/American Institute for Cancer Research (WCRF/AICR) have noted that dietary quality is a key factor influencing cancer risk, but most Americans do not meet these dietary guidelines for cancer prevention. The proposed study will enroll adults from the community (n=236 index participants, 236 household members; N = 472) who have low adherence to WCRF/AICR's four dietary guidelines. Participants will be randomized to either nutrition education or the Eatwell intervention. The Eatwell intervention content is focused on helping participants make healthier grocery shopping decisions, eat at home more often to take advantage of the optimal defaults present there, and learn how to navigate temptation when eating away from home. The findings will be relevant not only to the field of cancer prevention, but to the prevention of other diseases for which dietary quality is important.

DETAILED DESCRIPTION:
The purpose of this study is to test an intervention that is designed to facilitate adherence to the dietary guidelines for cancer prevention (i.e., increase in intake of fruits, vegetables, and whole grains, and decrease in intake of processed food, red and processed meat, and sugar sweetened beverages). Using a two-arm design, participants will be randomized to receive the "Eatwell" intervention or traditional nutrition education. The Eatwell intervention content is focused on helping participants make healthier grocery shopping decisions, eat at home more often to take advantage of the optimal defaults present there, and learn how to navigate temptation when eating away from home.

Aim 1: Test the hypothesis that there will be a greater increase in adherence to dietary guidelines for cancer prevention among index participants in the Eatwell condition, compared to the traditional nutrition condition. The primary outcome will be a total dietary adherence score, calculated using NCI's standardized scoring system. Grams per day of fruit, vegetables, and fiber; percentage of calorie intake from ultra-processed foods; grams per week of red meat and processed meat; and grams per day of SSBs will be examined individually as secondary outcomes.

Aim 2: Test the hypothesis that there will be greater improvements in biomarkers of inflammation among index participants in the Eatwell condition, compared to the traditional nutrition condition.

Aim 3: Test the hypothesis that adult household members will have greater improvements in dietary adherence (measured by total dietary adherence score, as well as change in individual components of dietary quality, as in Aim 1) when their index participant is randomized to the Eatwell condition, compared to the traditional nutrition condition.

Aim 4: Examine biopsychosocial mediators and moderators of intervention effects.

Aim 5: Exploratory analyses also will be conducted to, for example, examine change over time in the variables assessed as part of the study's assessment battery, understand predictors of change over time, and understand how independent or dependent variables are related to each other.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Access to technology necessary to receive emails and join videoconferencing meetings
* Ability to read and speak English
* Willingness to be randomized to either study condition, including ability and willingness to attend intervention sessions
* Ability and willingness to attend intervention sessions, receive monthly email messages, and serve in support role if index participant in household is assigned to Eatwell condition
* Able and willing to visit a commercial laboratory partnered with this project (e.g., Labcorp) in order to have their blood drawn at the time of study visits
* Low adherence to WCRF/AICR's four dietary guidelines (operationalized as a level of intake, based on brief self-report questions administered during phone screening, that corresponds to a score of 2 or less in the Shams-White method of dietary adherence scoring)
* Share a household (i.e., a private residence with a shared living space, including kitchen) with an adult who provides informed consent, meets eligibility criteria, and anticipates remaining in this household for the majority of the next 18 months
* Agree that they will not join another intervention study run by this study team in the next 18 months
* Successful completion by self and household member of all enrollment and baseline data collection tasks
* Have an email that they regularly check and willingness to use that for corresponding to study staff
* Weight at baseline of 396 lbs or less, as the digital scales used for measurement are not able to obtain measurements for weights higher than this

Exclusion Criteria:

* A medical or psychiatric condition, including self-reported history of anorexia nervosa or bulimia nervosa, that may limit appropriateness of or ability to comply with dietary recommendations
* A psychiatric condition, including self-reported history of anorexia nervosa or bulimia nervosa, that may make it difficult or inappropriate for household member to serve in support role
* Currently taking medication that can substantively change appetite or eating behavior, including using of a GLP-1 medication
* Planning to enroll in another lifestyle modification program in the next 18 months
* History of bariatric surgery
* Currently pregnant or planning to become pregnant in the next 18 months
* Type 1 Diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 472 (Estimated)
Dates: Start 2026-01-12 (Actual); Primary Completion 2029-11-30 (Estimated); Study Completion 2029-11-30 (Estimated)

PRIMARY OUTCOMES:
Total dietary adherence score | 0, 6, 18 months
  Index participants will complete the ASA24 for 2 weekdays and 1 weekend day at each assessment point. A research assistant (blind to study condition) will complete each food recall with the participant via videoconference, unless a participant indicates that they prefer to complete it independently. Information on dietary intake from the ASA24 will be used to calculate the total dietary adherence score, which is the primary outcome.

SECONDARY OUTCOMES:
Intake of targeted food groups | 0, 6, 18 months
  Index participants will complete the ASA24 for 2 weekdays and 1 weekend day at each assessment point. A research assistant (blind to study condition) will complete each food recall with the participant via videoconference, unless a participant indicates that they prefer to complete it independently. The data collected from the ASA24 will be used to examine change in intake of the individual components of the WCRF/AICR guidelines, including grams per day of fruit and vegetables, grams per day of fiber, percentage of calorie intake from ultra-processed foods, grams per week of red meat and processed meat, and grams per days or sugar sweetened drinks.
Inflammation | 0, 6, 18 months
  Inflammation will be measured, for index participants only, with two biomarkers. Interleukin-6 (IL-6) is a pleiotropic cytokine that plays an important role in the proliferation and differentiation of cells. C-reactive protein (CRP) is produced by the liver in response to circulating inflammatory mediators. CRP measurement will be done with high sensitivity analyses, which detect lower levels of protein than the standard assay. Participants will be asked not to engage in vigorous exercise or weightlifting in the 24 hours prior to the test.
Dietary quality | 0, 6, 18 months
  Index participants and their designated household members will each complete the Diet History Questionnaire-III (DHQ-III) once at each assessment point. The DHQ-III is a self-report survey that is completed online via an NCI website. This measure yields a total Healthy Eating Index-2015 (HEI-2015) score as well as specific subcomponents relevant to WCRF/AICR recommendations, such as added sugars.

OTHER OUTCOMES:
Participant age | 0 months
  Age at baseline will be self reported
Participant weight | 0 months
  Baseline weight will be self reported in pounds
Participant height | 0 months
  Height will be self reported in feet and inches
Participant race | 0 months
  Race will be self reported
Participant ethnicity | 0 months
  Ethnicity will be self reported
Participant gender | 0 months
  Gender will be self reported
Participant biological sex | 0 months
  Biological sex will be self reported
Participant household income | 0 months
  Household income at baseline will be self reported
Objectively measured weight | 0, 6, 18 months
  Each index participant will be provided with a Withings wireless scale, accurate to >0.2 kg, that transmits information directly to study staff. Scale information will be piped from the device to REDCap. Participants will be instructed to weigh themselves in the morning, after voiding urine but before eating, for three consecutive days at each assessment point, with the scale on a flat, hard surface. Data will be checked for outliers and averaged at each time point for each participant. BMI will be calculated based on self-reported height and objectively measured weight.
Physical Acitvity | 0, 6, 18 months
  Physical activity will be measured with the International Physical Activity Questionnaire.
Food insecurity | 0 months
  This will be assessed with the USDA's Household Food Security Survey and will be dichotomized as food secure vs. low or very low security.
Neighborhood food environment | 0 months
  The neighborhood food environment will be assessed through the use of the modified Retail Food Environment Index (mRFEI) score, sourced from the CDC and census tract. Participant addresses will be used to determine their mRFEI score.
The proportion of meals and snacks sourced from grocery stores | 0, 6, 18 months
  This will be measured with the "Source" module on ASA24 food recalls, which tags each food entry with a source (e.g., convenience store, fast food, street vendor, etc.). Participants will be categorized into tertiles based on proportion of diet sourced from grocery stores.
Treatment Acceptability | 6, 18 months
  Treatment Acceptability will be measured at 6 and 18 months using the Treatment Acceptability Questionnaire. This measure was created by the study team.
Self-regulation | 0, 6, 18 months
  To measure use of self-regulation strategies, participants will be asked to rate the frequency with which they used each strategy in the past month. Change in use of intervention-targeted strategies will be examined.
Self-regulation | 0, 6, 18 months
  Self-regulation will also be measured through the Power of Food Scale.
Autonomous Motivation | 0, 6, 18 months
  Autonomous motivation for dietary change will be examined with the Treatment Self-Regulation Questionnaire.
Supportive Accounability | 0, 6, 18 months
  Supportive accountability will be measured with the dietary items of the Supportive Accountability Measure.
Social Support | 0, 6, 18 months
  Social support for healthy eating from household members will be measured with select items adapted from Sallis's Social Support for Diet Survey and the Quality of Interactions survey.

CONTACTS AND LOCATIONS:
Locations (1):
- Drexel University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
All deidentified data will be placed in a public repository.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Within 12 months after study completion.
Access Criteria: Public availability
URL: https://drexel.edu/coas/faculty-research/faculty-directory/psychology-well/faculty-core/Meghan-Butryn/